CLINICAL TRIAL: NCT01178333
Title: Heparin-Induced Thrombocytopenia - Retrospective Analysis of Data on Incidence and Outcomes Study (HIT-RADIO Study)
Brief Title: Heparin-Induced Thrombocytopenia - Retrospective Analysis of Data on Incidence and Outcomes Study
Acronym: HIT-RADIO
Status: Completed | Type: Observational
Sponsor: Carelon Research (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 678; U01HL072268 (NIH)
Record Dates: First submitted 2010-08-06; First posted 2010-08-10 (Estimated); Results first posted 2015-05-04 (Estimated); Last update posted 2015-05-22 (Estimated); Status verified 2013-03

CONDITIONS: Heparin Induced Thrombocytopenia
Keywords: Thrombocytopenia; Heparin
MeSH Terms: conditions — Thrombocytopenia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
HIT-RADIO is a study of patients who had a positive heparin PF-4 antibody test between 1/21/2008 and 9/25/2008 at selected hospitals. The study will collect and analyse information that is already in the patients' medical records. Information about laboratory values (such as platelet counts), treatments (such as medications), and outcomes (such as blood clots, amputation, and death) will be included.

DETAILED DESCRIPTION:
HIT-RADIO is a retrospective chart-review study of patients who had a positive heparin PF-4 antibody test between 1/21/2008 and 9/25/2008 at selected hospitals associated with the Transfusion Medicine/Hemostasis Clinical Trials Network .

Heparin-induced thrombocytopenia (HIT) is a major complication of the administration of heparin and can result in life-threatening thrombosis with or without thrombocytopenia (HIT-T) or can produce thrombocytopenia without clinically symptomatic thrombosis ("isolated" HIT). Isolated heparin-induced thrombocytopenia is defined as a fall in platelet count associated with a positive heparin PF-4 antibody test, in the absence of clinically overt thrombosis. While the treatment of HIT-T (HIT with thrombosis) with anticoagulation is well established, the risks and treatment of isolated HIT are unclear.

It is anticipated that this data analysis will provide a current overview of the implications of a positive heparin PF-4 antibody test in clinical practice. It should determine the percentage of positive heparin PF-4 antibody tests that are associated with thrombocytopenia and thrombosis (HIT-T) or "isolated" HIT at diagnosis and the subsequent major clinical outcomes of death, limb amputation/gangrene, and new thrombosis. No "snapshot" of such HIT patients has been conducted in the past decade and the results will be important in assessing the impact of HIT in current medical care as well as documenting current treatment strategies.

ELIGIBILITY:
Inclusion Criteria:

* All subjects with a positive heparin PF-4 antibody test occurring between 1/21/2008 and 9/25/2008
* Medical record available for the admission during which the positive heparin PF-4 antibody test was obtained

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects with a positive heparin PF-4 antibody test drawn between 1/21/2008 and 9/25/2008
Sampling Method: Probability Sample
Enrollment: 668 (Actual)
Dates: Start 2010-06; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan F Assmann, PhD, Principal Investigator — Carelon Research; David Kuter, MD, Principal Investigator — Massachusetts General Hospital; Eliot Williams, MD PHD, Principal Investigator — University of Wisconsin, Madison; Kenneth Friedman, MD, Principal Investigator — Versiti Blood Health; Ronald Go, MD, Principal Investigator — Gunderson Clinic; Keith McCrae, MD, Principal Investigator — The Cleveland Clinic; Ellis Neufeld, MD PHD, Principal Investigator — Boston Children's Hospital; Lynne Uhl, MD, Principal Investigator — Beth Israel Deaconess Medical Center; Judith Lin, MD, Principal Investigator — Brigham and Women's Hospital; James Bussel, MD, Principal Investigator — Cornell University; Thomas Ortel, MD PHD, Principal Investigator — Duke University; Jodi Segal, MD MPH, Principal Investigator — Johns Hopkins University; Barbara Konkle, MD, Principal Investigator — Bloodworks; Cindy Leissinger, MD, Principal Investigator — Tulane University; Thomas Raife, MD, Principal Investigator — University of Iowa; Ann Zimrin, MD, Principal Investigator — University of Maryland Greenebaum Cancer Center; Jeffrey McCullough, MD, Principal Investigator — University of Minnesota; Nigel Key, MD, Principal Investigator — University of North Carolina, Chapel Hill; Bruce Sachais, MD PHD, Principal Investigator — University of Pennsylvania; Joseph Kiss, MD, Principal Investigator — University of Pittsburgh Institute for Transfusion Medicine
Locations (21):
- United States (21):
  - University of Iowa, Iowa City, Iowa
  - Tulane University, New Orleans, Louisiana
  - University of Maryland Greenebaum Cancer Center, Baltimore, Maryland
  - Johns Hopkins, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Children's Hospital, Boston, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - University of Minnesota, Minneapolis, Minnesota
  - Cornell University, New York, New York
  - University of North Carolina, Chapel Hill, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Case Western Reserve University School of Medicine, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Gunderson Clinic, La Crosse, Wisconsin
  - University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin
  - Froedtert, Milwaukee, Wisconsin
  - St. Luke's Medical Center, Milwaukee, Wisconsin

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Of 668 consecutive patients with a positive heparin-PF4 ELISA test, 226 were excluded, primarily due to lack of recent heparin exposure. Of 442 eligible patients, 71 had HIT-T, 284 had Isolated HIT and 87 had no HIT.
Groups:
- HIT-T: Positive heparin-PF4 ELISA test and a thrombotic event associated with heparin exposure within the preceding 5 days (and with the onset of a platelet count drop of >15% beginning within 5-10 days after starting heparin), with or without thrombocytopenia.
- Isolated HIT: Positive heparin-PF4 ELISA test and a nadir platelet count <50% of baseline platelet count associated with heparin exposure in the preceding 5 days (and with the onset of a platelet count drop of >15% beginning within 5-10 days after starting heparin), without a thrombotic event.
- No HIT: Positive heparin-PF4 ELISA test with heparin exposure in the preceding 5 days, but not meeting criteria for HIT-T or isolated HIT.
Period: Overall Study
Arm/Group | HIT-T | Isolated HIT | No HIT
Started | 71 | 284 | 87
Completed | 71 | 284 | 87
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Of 668 consecutive patients with a positive heparin-PF4 ELISA test, 225 were excluded, primarily due to lack of recent heparin exposure. Of 442 eligible patients, 71 had HIT-T, 284 had Isolated HIT and 87 had no HIT.
Groups:
- Total: Total of all reporting groups
Arm/Group | HIT-T | Isolated HIT | No HIT | Total
Number analyzed (Participants) | 71 | 284 | 87 | 442
Age, Continuous [Mean (Standard Deviation); unit: years] | 62 (16) | 59 (18) | 60 (19) | 60 (18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 144 | 40 | 223
  Male | 32 | 140 | 47 | 219
Baseline Platelet Count [Mean (Standard Deviation); unit: x 10^9/L] | 282 (268) | 270 (149) | 215 (172) | 261 (158)
Heparin exposure this admission before Day 0: use (or non-use) of unfractionated heparin (UFH) [Number; unit: participants] — Two types of heparins are commonly used as anticoagulants - unfractionated heparin (UFH) and low-molecular-weight heparin (LMWH). Unfractionated heparin (UFH) has been used for the prevention and treatment of thrombosis for several decades.
  participants
    Use of unfractionated heparin | 67 | 263 | 79 | 409
    Non-use of unfractionated heparin | 4 | 21 | 8 | 33
Heparin exposure this admission before Day 0: use (or non-use) of low molecular weight heparin [Number; unit: participants] — Two types of heparins are commonly used as anticoagulants - unfractionated heparin (UFH) and low-molecular-weight heparin (LMWH). Low molecular weight heparin (LMWH) is derived from UFH by depolymerization. Each LMWH product has a specific molecular weight distribution that determines its anticoagulant activity and duration of action.
  participants
    Use of low molecular weight heparin | 15 | 48 | 11 | 74
    Non-use of low molecular weight heparin | 56 | 236 | 76 | 368
Heparin-PF4 (platelet factor 4) OD (optical density) test results [Number; unit: participants] — The OD in the Heparin-PF4 OD test stands for optical density. The PF4 stands for platelet factor 4. The test looks for antibodies to complexes of heparin combined with platelet factor 4. Higher optical density indicates higher antibody concentration. We could say that generally OD values above 0.4 are considered a positive result, and that the higher the OD, the greater the concentration of antibodies in the patient's blood.
  participants
    Less than 1.0 | 34 | 163 | 61 | 258
    Greater than or equal to 1.0 | 37 | 120 | 26 | 183
    Missing | 0 | 1 | 0 | 1
Admitting service [Number; unit: participants]
  CV/thoracic surgery | 18 | 78 | 18 | 114
  Orthopedic surgery | 2 | 9 | 4 | 15
  Other surgery | 15 | 33 | 8 | 56
  Medicine | 36 | 161 | 56 | 253
  Missing | 0 | 3 | 1 | 4

OUTCOME MEASURES:

1. Secondary Outcome: Time to Death
Description: The mean time to an event is estimated by the area under the survival function. If the largest time is an event time, then the survival function goes to zero at that time, and the mean survival estimate is finite. Otherwise, the mean time cannot be estimated and may lead to a bias.
Time Frame: From the time the positive heparin PF-4 antibody test was drawn until hospital discharge, death, or day 45, whichever occurred first
Measure: Mean (Standard Error); unit: days
Arm/Group | HIT-T | Isolated HIT | No HIT
Number analyzed (Participants) | 71 | 284 | 87
days | 23.6 (1.43) | 35.4 (1.11) | 34.5 (2.64)
Statistical Analysis 1: Comparison: HIT-T vs No HIT; Test type: Superiority or Other; p = 0.09, Regression, Cox; Hazard Ratio (HR) = 1.98, 95% CI 2-sided [0.90 to 4.36]
Statistical Analysis 2: Comparison: Isolated HIT vs No HIT; Test type: Superiority or Other; p = 0.45, Regression, Cox; Hazard Ratio (HR) = 1.31, 95% CI 2-sided [0.65 to 2.66]

2. Secondary Outcome: Time to Death
Description: The median survival time is reported by each group for the time to death.
Time Frame: as for outcome 1
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | HIT-T | Isolated HIT | No HIT
Number analyzed (Participants) | 71 | 284 | 87
days | 31.0 [23.0 to NA] — Due to lack of events, the upper interval of the median survival time could not be estimated. | NA [NA to NA] — Due to lack of events, the median survival time and 95% confidence interval could not be estimated. | NA [29.0 to NA] — Due to lack of events, the median survival time and the upper interval could not be estimated.

3. Secondary Outcome: Time to Occurrence of Limb Amputation or Limb Gangrene
Description: Due to the small number of events, the median or mean survival time could not be defined. Therefore, the number of subjects with limb amputation or limb gangrene was reported in "Outcome Measure Data Table".
Time Frame: as for outcome 1
Measure: Number; unit: participants
Arm/Group | HIT-T | Isolated HIT | No HIT
Number analyzed (Participants) | 71 | 284 | 87
participants | 5 | 6 | 1
Statistical Analysis 1: Comparison: HIT-T vs No HIT; Test type: Superiority or Other; p = 0.15, Regression, Cox; Hazard Ratio (HR) = 4.76, 95% CI 2-sided [0.55 to 40.87]
Statistical Analysis 2: Comparison: Isolated HIT vs No HIT; Test type: Superiority or Other; p = 0.78, Regression, Cox; Hazard Ratio (HR) = 1.35, 95% CI 2-sided [0.16 to 11.25]

4. Secondary Outcome: Time to Occurrence of Radiographically Confirmed Thromboembolism
Description: The mean time to an event is estimated by the area under the survival function. If the largest time is an event time, then the survival function goes to zero at that time, and the mean survival estimate is finite. Otherwise, the mean time cannot be estimated and may lead to a bias. However, the median survival times could not be defined for all three groups, so the mean time was reported in "Outcome Measure Data Table".
Time Frame: as for outcome 1
Measure: Mean (Standard Error); unit: days
Arm/Group | HIT-T | Isolated HIT | No HIT
Number analyzed (Participants) | 71 | 284 | 87
days | 11.1 (0.48) | 26.1 (0.74) | 5.74 (0.11)
Statistical Analysis 1: Comparison: HIT-T vs No HIT; Test type: Superiority or Other; p = 0.06, Regression, Cox; Hazard Ratio (HR) = 2.38, 95% CI 2-sided [0.98 to 5.79]
Statistical Analysis 2: Comparison: Isolated HIT vs No HIT; Test type: Superiority or Other; p = 0.11, Regression, Cox; Hazard Ratio (HR) = 1.91, 95% CI 2-sided [0.87 to 4.21]

5. Secondary Outcome: Time to Occurrence of Major Bleeding
Description: as for outcome 1
Time Frame: From the time that the positive heparin PF-4 antibody test was drawn until hospital discharge, death, or day 45, whichever occurred first
Measure: Mean (Standard Error); unit: days
Arm/Group | HIT-T | Isolated HIT | No HIT
Number analyzed (Participants) | 71 | 284 | 87
days | 15.6 (1.54) | 26.5 (1.36) | 17.2 (0.97)
Statistical Analysis 1: Comparison: HIT-T vs No HIT; Test type: Superiority or Other; p = 0.001, Regression, Cox; Hazard Ratio (HR) = 2.80, 95% CI 2-sided [1.50 to 5.22]
Statistical Analysis 2: Comparison: Isolated HIT vs No HIT; Test type: Superiority or Other; p = 0.02, Regression, Cox; Hazard Ratio (HR) = 1.97, 95% CI 2-sided [1.12 to 3.45]

6. Secondary Outcome: Time to Occurrence of Major Bleeding
Description: The median survival time is reported by each group for the time to occurrence of major bleeding.
Time Frame: as for outcome 5
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | HIT-T | Isolated HIT | No HIT
Number analyzed (Participants) | 71 | 284 | 87
days | 17.0 [8.0 to 28.0] | 36.0 [31.0 to NA] — Due to lack of events, the upper interval of median survival time could not be estimated. | NA [16.0 to NA] — Due to lack of events, the median survival time and the upper interval could not be estimated.

7. Secondary Outcome: Proportion of Subjects With HIT With Thrombosis (HIT-T) and Isolated HIT
Description: Proportion of subjects who, at the time the positive heparin PF-4 antibody test was drawn, were in each of the following categories:
  * Group 1: Those with thrombosis and or without thrombocytopenia (HIT-T): 16% of 442 subjects.
  * Group 2: Those with thrombocytopenia but not thrombosis (Isolated HIT): 64% of 442 subjects.
  * Group 3: Those with neither thrombocytopenia nor thrombosis (Neither HIT-T nor Isolated HIT): 20% of 442 subjects.
Time Frame: From the date 5 days before the positive heparin PF-4 antibody test was drawn to the date it was drawn
Measure: Number; unit: participants
Arm/Group | HIT-T | Isolated HIT | No HIT
Number analyzed (Participants) | 71 | 284 | 87
participants | 71 | 284 | 87

8. Secondary Outcome: Type of Heparin Exposure - Unfractionated Heparin (UFH)
Description: Two types of heparins are commonly used as anticoagulants - unfractionated heparin (UFH) and low-molecular-weight heparin (LMWH). UFH has been used for the prevention and treatment of thrombosis for several decades.
Time Frame: Hospital admission to date the positive heparin PF-4 antibody test was drawn, or 28 days prior to the date it was drawn, whichever is later, through the date it was drawn
Measure: Number; unit: participants
Arm/Group | HIT-T | Isolated HIT | No HIT
Number analyzed (Participants) | 71 | 284 | 87
participants
  Number of subjects with heparin exposure:UFH | 67 | 263 | 79
  Number of subjects without heparin exposure:UFH | 4 | 21 | 8
Statistical Analysis 1: Comparison: HIT-T vs Isolated HIT vs No HIT; Test type: Superiority or Other; p = 0.72, Chi-squared — P-value is to compare three groups

9. Secondary Outcome: Type of Heparin Exposure - Low Molecular Weight Heparin (LMWH)
Description: Two types of heparins are commonly used as anticoagulants - unfractionated heparin (UFH) and low-molecular-weight heparin (LMWH). LMWHs are derived from UFH by depolymerization. Each LMWH product has a specific molecular weight distribution that determines its anticoagulant activity and duration of action.
Time Frame: as for outcome 8
Measure: Number; unit: participants
Arm/Group | HIT-T | Isolated HIT | No HIT
Number analyzed (Participants) | 71 | 284 | 87
participants
  Number of subjects with heparin exposure:LMWH | 15 | 48 | 11
  Number of subjects without heparin exposure:LMWH | 56 | 236 | 76
Statistical Analysis 1: Comparison: HIT-T vs Isolated HIT vs No HIT; Test type: Superiority or Other; p = 0.37, Chi-squared — P-value is to compare three groups

10. Secondary Outcome: Relationship of the Heparin PF-4 (Platelet Factor 4) Antibody Titer to the Clinical Diagnosis
Description: Heparin PF-4 (platelet factor 4) optical density (OD) test results were the dichotomous outcome (<1.0 vs. >=1.0). Clinical diagnosis was three groups (HIT-T, Isolated HIT and No HIT). The Heparin PF-4 optical density test looks for antibodies to complexes of heparin combined with platelet factor 4. Higher optical density indicates higher antibody concentration. We could say that generally OD values above 0.4 are considered a positive result, and that the higher the OD, the greater the concentration of antibodies in the patient's blood.
Time Frame: as for outcome 1
Population: There was one missing data for optical density test results in Isolated HIT group. Therefore, 283 subjects were used for Isolated HIT group.
Measure: Number; unit: participants
Arm/Group | HIT-T | Isolated HIT | No HIT
Number analyzed (Participants) | 71 | 283 | 87
participants
  Optical density Results less than 1.0 | 34 | 163 | 61
  Optical density Results greater or equal to 1.0 | 37 | 120 | 26
Statistical Analysis 1: Comparison: HIT-T vs Isolated HIT vs No HIT; Test type: Superiority or Other; p = 0.02, Chi-squared — P-value is to compare three groups

11. Secondary Outcome: Relationship of the Heparin PF-4 Antibody Titer to the Degree of Thrombocytopenia
Description: Heparin PF-4 optical density (OD) test results were the dichotomous outcome (<1.0 vs. >=1.0). Nadir Platelet Count (x10^9 / L) was used for the degree of thrombocytopenia. The Heparin PF-4 optical density test looks for antibodies to complexes of heparin combined with platelet factor 4. Higher optical density indicates higher antibody concentration. We could say that generally OD values above 0.4 are considered a positive result, and that the higher the OD, the greater the concentration of antibodies in the patient's blood.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: X10^9 / L
Groups:
- OD Result < 1.0: Heparin-PF4 OD Test Results < 1.0
- OD Result >= 1.0: Heparin-PF4 OD Test Results >= 1.0
Arm/Group | OD Result < 1.0 | OD Result >= 1.0
Number analyzed (Participants) | 258 | 183
X10^9 / L | 87.7 (92.4) | 83.1 (76.4)
Statistical Analysis 1: Comparison: OD Result < 1.0 vs OD Result >= 1.0; Test type: Superiority or Other; p = 0.58, ANOVA

12. Secondary Outcome: Relationship of the Heparin PF-4 Antibody Titer to the Primary Endpoint
Description: Heparin PF-4 OD test results were the dichotomous outcome (<1.0 vs. >=1.0). Primary endpoint was the composite endpoint of death, limb amputation/gangrene, or new thrombosis.
Time Frame: as for outcome 1
Measure: Number; unit: participants
Arm/Group | OD Result < 1.0 | OD Result >= 1.0
Number analyzed (Participants) | 258 | 183
participants
  Composite endpoint | 85 | 66
  No composite endpoint | 173 | 117
Statistical Analysis 1: Comparison: OD Result < 1.0 vs OD Result >= 1.0; Test type: Superiority or Other; p = 0.66, Regression, Cox

13. Secondary Outcome: Use of Treatment (Non-heparin Anticoagulant) Used in Hospital
Description: Types of treatment (direct thrombin inhibitor, fondaparinux, warfarin, no treatment) provided to subjects in hospital
Time Frame: as for outcome 5
Measure: Number; unit: participants
Arm/Group | HIT-T | Isolated HIT | No HIT
Number analyzed (Participants) | 71 | 284 | 87
participants
  Number of subjects with treatment in hospital | 58 | 167 | 43
  Number of subjects without treatment in hospital | 13 | 117 | 44
Statistical Analysis 1: Comparison: HIT-T vs Isolated HIT vs No HIT; Test type: Superiority or Other; p < 0.01, Chi-squared — P-value is to compare three groups

14. Primary Outcome: Time to Occurrence of a Composite Triple Endpoint Consisting of Death, Limb Amputation/Gangrene, and New Thrombosis
Description: as for outcome 1
Time Frame: From the time that the positive heparin PF-4 antibody test was drawn until hospital discharge or day 45, whichever occurred first.
Measure: Mean (Standard Error); unit: days
Arm/Group | HIT-T | Isolated HIT | No HIT
Number analyzed (Participants) | 71 | 284 | 87
days | 17.5 (1.66) | 27.8 (1.30) | 31.4 (2.67)
Statistical Analysis 1: Comparison: HIT-T vs No HIT; Test type: Superiority or Other; p = 0.003, Regression, Cox; Hazard Ratio (HR) = 2.48, 95% CI 2-sided [1.35 to 4.55]
Statistical Analysis 2: Comparison: Isolated HIT vs No HIT; Test type: Superiority or Other; p = 0.07, Regression, Cox; Hazard Ratio (HR) = 1.66, 95% CI 2-sided [0.96 to 2.85]

15. Primary Outcome: Time to Occurrence of a Composite Triple Endpoint Consisting of Death, Limb Amputation/Gangrene, and New Thrombosis
Description: The median survival time is reported by each group for the time to occurrence of a composite triple endpoint consisting of death, limb amputation/gangrene, and new thrombosis.
Time Frame: as for outcome 14
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | HIT-T | Isolated HIT | No HIT
Number analyzed (Participants) | 71 | 284 | 87
days | 13.0 [9.0 to NA] — Due to lack of events, the upper interval of the median survival time could not be estimated. | 33.0 [25.0 to NA] — Due to lack of events, the upper interval of the median survival time could not be estimated. | NA [29.0 to NA] — Due to lack of events, the median survival time and the upper interval could not be estimated.

16. Secondary Outcome: Use of Treatment (Non-heparin Anticoagulant) Used at the Time of Discharge
Time Frame: as for outcome 5
Measure: Number; unit: participants
Arm/Group | HIT-T | Isolated HIT | No HIT
Number analyzed (Participants) | 71 | 284 | 87
participants
  Number of subjects with treatment at discharge | 57 | 159 | 39
  Number of subjects with no treatment at discharge | 14 | 125 | 48
Statistical Analysis 1: Comparison: HIT-T vs Isolated HIT vs No HIT; Test type: Superiority or Other; p < 0.01, Chi-squared — P-value is to compare three groups

17. Secondary Outcome: Time to Platelet Recovery, Among Subjects With a Low Platelet Count When the Positive PF4 Antibody Test Was Drawn
Time Frame: From the time that the nadir platelet count was drawn until hospital discharge, death, or day 45, whichever occurred first
Measure: Mean (Standard Error); unit: days
Arm/Group | HIT-T | Isolated HIT | No HIT
Number analyzed (Participants) | 52 | 249 | 40
days | 5.16 (0.92) | 5.16 (0.38) | 2.96 (0.33)
Statistical Analysis 1: Comparison: HIT-T vs No HIT; Test type: Superiority or Other; p = 0.72, Regression, Cox; Hazard Ratio (HR) = 0.92, 95% CI 2-sided [0.56 to 1.49]
Statistical Analysis 2: Comparison: Isolated HIT vs No HIT; Test type: Superiority or Other; p = 0.34, Regression, Cox; Hazard Ratio (HR) = 0.82, 95% CI 2-sided [0.54 to 1.24]

ADVERSE EVENTS:
Description: HIT-RADIO was a retrospective study so there were no adverse events collected/reported.
Arm/Group | HIT-T | Isolated HIT | No HIT
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All publications and presentations resulting from studies from the TMH Network must be approved by the Publications and Presentations Committee before submission. The Sponsor (NERI) and funding agency (NHLBI) both are represented on the P&P Committee along with Network Investigators. Members of the P&P Committee can recommend changes to publications.